CLINICAL TRIAL: NCT01565798
Title: Copper Antimicrobial Research Program: Environmental and Patient Sampling For Indicator Organisms To Determine The Efficacy Of Copper To Reduce Acquisition Of Microbes From The Patient Care Environment
Brief Title: Efficacy Of Copper To Reduce Acquisition Of Microbes and Healthcare-acquired Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other); Ralph H. Johnson VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: DOD W81XWH-07-C-0053; Effect of Copper on HAI (Other Grant/Funding Number: U.S. Army Material Command Contract W81XWH-07-C-0053)
Record Dates: First submitted 2012-03-26; First posted 2012-03-29 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2011-12

CONDITIONS: Healthcare-acquired Infection
Keywords: healthcare-acquired infections; colonization; copper-alloy surfaces

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Copper Surfaced Room (Experimental): Patients sequentially randomized to this arm were admitted to an ICU room with copper surfaced objects.
  Interventions: Other: Copper-alloy surfaced patient care objects
- Standard Surfaced Room (No Intervention): Patients sequentially randomized to this arm were admitted to an ICU room with standard surfaced objects

INTERVENTIONS:
Other: Copper-alloy surfaced patient care objects — Copper-alloy surfaced bed rails, over bed tray tables, chair arms, nurse call devices, laptop and computer monitor bezels, and IV poles were placed into the patient ICU rooms.
  Arms: Copper Surfaced Room

SUMMARY:
CONTEXT: Healthcare-acquired infections (HAI) cause substantial patient morbidity and mortality. Commonly touched items in the patient care environment harbor microorganisms that may contribute to HAI risk. Thus, reduction in the surface bioburden may be an effective strategy to reduce HAI. Inherent biocidal capabilities of copper surfaces offer a theoretical advantage to conventional cleaning, as disinfection is continuous rather than episodic.

OBJECTIVE: Determine whether placement of copper-alloy surfaced objects in an intensive care unit (ICU) reduce risk of HAI.

DESIGN: An intention to treat study where patients are sequentially placed into rooms with or without copper-alloy surfaced objects.

SETTING: The ICUs of three hospitals, a tertiary academic hospital, an academic cancer center, and a Veteran's Administration Medical Center.

PATIENTS: Any patient 18 years of age or older who required admission to an ICU at a study hospital is eligible for placement into a study room if available.

INTERVENTION: Placement of copper-alloy surfaced objects in an ICU room. MAIN OUTCOME MEASURE: Rate of incident HAI and/or colonization with methicillin-resistant Staphylococcus aureus (MRSA) or vancomycin-resistant Enterococcus (VRE) in each type of room.

ELIGIBILITY:
Inclusion Criteria:

patients 18 years and older requiring admission to an ICU at one of the study sites were eligible

Exclusion Criteria:

* less than 18 years of age or
* pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2010-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Rate of incident HAI and/or colonization with methicillin-resistant Staphylococcus aureus (MRSA) or vancomycin-resistant Enterococcus (VRE) in each type of room. | July 2010 to June 2011 (up to 1 year)
  Patients prospectively followed from ICU admission to hospital discharge for acquisition of HAI and/or colonization with MRSA or VRE

SECONDARY OUTCOMES:
Microbial burden and risk of HAI | July 2010 to June 2011 (up to 1 year)
  The risk of HAI among patients admitted to ICU will be assessed by microbial burden of environment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael G Schmidt, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States